CLINICAL TRIAL: NCT01599689
Title: Can an Evidence-based Mirrors Intervention Reduce Postoperative Delirium in Older Cardiac Surgical Patients? A Pilot and Feasibility Cluster Randomised Controlled Trial
Brief Title: Pilot and Feasibility Study of a Mirrors Intervention for Reducing Delirium in Older Cardiac Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P01629; SA16/0212 (Other Grant/Funding Number: The Dunhill Medical Trust)
Record Dates: First submitted 2012-05-08; First posted 2012-05-16 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Delirium
Keywords: Delirium; Delirium, Dementia, Amnestic, Cognitive Disorders; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms; Mental Disorders; Cardiac Surgery; Mirrors
MeSH Terms: conditions — Emergence Delirium; Delirium; Neurocognitive Disorders; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirrors Intervention (Experimental): Patients allocated to Mirrors will receive a structured, protocol-driven bedside mirrors intervention as part of their postsurgical ICU care. This intervention will commence as soon as all anaesthetic agents have been switched off and the patient is awake following surgery unless considered clinically inappropriate.
  Interventions: Other: Mirrors Intervention
- Standard Care (No Intervention): Patients allocated to Standard Care will receive the usual postsurgical ICU care that does not include the use of mirrors.

INTERVENTIONS:
Other: Mirrors Intervention — Coaching in the use of two types of mirrors to support mental status and attention, physical mobility, and sense of body awareness and ownership, as well as patient dignity and privacy in self-care.
  To be administered at set times and in a standardised way by ICU nursing and physical therapy teams.
  Arms: Mirrors Intervention

SUMMARY:
This pilot cluster-randomised controlled trial aims to determine whether the use of bedside mirrors, as a clearly defined part of patients' postsurgical ICU care, can reduce delirium and improve outcomes in the older cardiac surgical patient.

DETAILED DESCRIPTION:
The risk of delirium, an acute disturbance in mental status and cognition that occurs commonly after cardiac surgery, increases sharply from the age of about 65 years. Its occurrence, even for one day, is associated with longer ICU and hospital stays, increased costs, and negative physical and cognitive outcomes at one year. In spite of previous prevention and intervention research, delirium incidence in the older cardiac surgical patient remains high (up to 72%).

ICU clinicians at Papworth Hospital have made observations suggesting that delirium could be reduced using a novel and unconventional strategy of bedside mirrors. Mirrors of any type are uncommon in ICU environments[1], but their occasional use by patients on our ICU has been reported by bedside clinicians and physiotherapists to result in:

* a normalisation of mental status and attention (core delirium diagnostic criteria), and
* earlier physical mobilisation (associated with reduced delirium risk), particularly in older-aged patients

Evidence from other sources supports mirrors' beneficial effect in these areas [2-10], but mirror use has never to our knowledge been explored for the reduction of delirium. This pilot study seeks to determine whether the use of bedside mirrors, as a clearly defined part of patients' postsurgical ICU care, can reduce delirium and improve outcomes in the older cardiac surgical patient.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective or urgent cardiac surgery at Papworth Hospital
* aged 70+ years

Exclusion Criteria:

* inability to obtain informed consent
* care pathway anticipating admission elsewhere than to ICU following surgery
* severe visual impairment impeding ability to recognise self in mirror
* physical or communication barriers likely to impede effective administration of study procedures
* severe mental disability likely to impede effective administration of study procedures or assessment of delirium
* history of psychiatric illness previously requiring hospitalisation

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Delirium incidence | Assessed from day of ICU admission after surgery until day of ICU discharge (or until 12 weeks after surgery, whichever comes first)
  Delirium will be measured twice daily, using the Confusion Assessment Method for the ICU (CAM-ICU).

SECONDARY OUTCOMES:
Delirium time of onset | Assessed from day of ICU admission after surgery until day of ICU discharge (or until 12 weeks after surgery, whichever comes first)
  This is the patient's first occurrence of delirium, as measured using the CAM-ICU, counted in number of days from admission to ICU.
Delirium duration | Assessed from day of ICU admission after surgery until day of ICU discharge (or until 12 weeks after surgery, whichever comes first)
  This is the total number of ICU days with delirium, as measured using the CAM-ICU
Mental Status | Assessed from day of ICU admission after surgery until day of ICU discharge (or until 12 weeks after surgery, whichever comes first)
  Measured from Features 1 & 3 of CAM-ICU
Attention | Assessed from day of ICU admission after surgery until day of ICU discharge (or until 12 weeks after surgery, whichever comes first)
  Measured from Feature 2 of CAM-ICU
Functional Independence | Assessed at 12 weeks after surgery
  Measured using Barthel Index
Perceptual disturbances about the body and dissociative symptoms | Assessed at 12 weeks after surgery
  Measured using interview described in previous work (Morgan et al., Biol Psychiatry, 2011)
Health-Related Quality of Life (HRQoL) | Assessed at 12 weeks after surgery
  Measured using EQ-5D
Length of ICU and hospital stay | Assessed at hospital hospital discharge
  This is the patient's length of stay in ICU and hospital, in number of days from admission date until discharge date.
Mortality | Assessed at 12 weeks after surgery
  This is patient mortality from admission to ICU until 12 weeks after surgery.
Factual memories from ICU | Assessed at 12 weeks after surgery
  Measured using the ICU Memory Tool (Jones et al., Clin Intensive Care, 2000)
Intraclass correlation coefficient (ICC) for time clusters | Assessed from day of ICU admission after surgery until day of ICU discharge (or until 12 weeks after surgery, whichever comes first)
  This is a measure of the within-cluster correlation necessary for calculating sample size necessary for a definitive trial if warranted
Acceptability of the intervention | Assessed from day of ICU admission after surgery until day of ICU discharge (or until 12 weeks after surgery, whichever comes first)
  This is the number of instances when the intervention was considered appropriate by clinicians and accepted and used by patients, divided by total recorded indicated instances.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alain Vuylsteke, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Freysteinson WM. The use of mirrors in critical care nursing. Crit Care Nurs Q. 2009 Apr-Jun;32(2):89-93. doi: 10.1097/CNQ.0b013e3181a27b3d. PMID 19300071
- [Background] Vanhaudenhuyse A, Schnakers C, Bredart S, Laureys S. Assessment of visual pursuit in post-comatose states: use a mirror. J Neurol Neurosurg Psychiatry. 2008 Feb;79(2):223. doi: 10.1136/jnnp.2007.121624. No abstract available. PMID 18202215
- [Background] Tabak N, Bergman R, Alpert R. The mirror as a therapeutic tool for patients with dementia. Int J Nurs Pract. 1996 Sep;2(3):155-9. doi: 10.1111/j.1440-172x.1996.tb00042.x. PMID 9265610
- [Background] Altschuler EL, Wisdom SB, Stone L, Foster C, Galasko D, Llewellyn DM, Ramachandran VS. Rehabilitation of hemiparesis after stroke with a mirror. Lancet. 1999 Jun 12;353(9169):2035-6. doi: 10.1016/s0140-6736(99)00920-4. No abstract available. PMID 10376620
- [Background] Tung ML, Murphy IC, Griffin SC, Alphonso AL, Hussey-Anderson L, Hughes KE, Weeks SR, Merritt V, Yetto JM, Pasquina PF, Tsao JW. Observation of limb movements reduces phantom limb pain in bilateral amputees. Ann Clin Transl Neurol. 2014 Sep;1(9):633-8. doi: 10.1002/acn3.89. Epub 2014 Sep 30. PMID 25493277
- [Derived] Giraud K, Pontin M, Sharples LD, Fletcher P, Dalgleish T, Eden A, Jenkins DP, Vuylsteke A. Use of a Structured Mirrors Intervention Does Not Reduce Delirium Incidence But May Improve Factual Memory Encoding in Cardiac Surgical ICU Patients Aged Over 70 Years: A Pilot Time-Cluster Randomized Controlled Trial. Front Aging Neurosci. 2016 Sep 28;8:228. doi: 10.3389/fnagi.2016.00228. eCollection 2016. PMID 27733826